CLINICAL TRIAL: NCT01144806
Title: Evaluation of Energy Expenditure, Body Composition and Recovery Rates in Children With Severe Acute Malnutrition (SAM) Receiving Community-based Nutritional Rehabilitation Therapy
Brief Title: Evaluation of Energy Expenditure, Body Composition and Recovery Rates in Children With Severe Acute Malnutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: International Atomic Energy Agency (Other Government)
Responsible Party: Principal Investigator, Dr Zulfiqar Ahmed Bhutta, Principal Investigator, Aga Khan University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1400-Ped-ERC-09
Record Dates: First submitted 2010-06-15; First posted 2010-06-16 (Estimated); Last update posted 2012-02-27 (Estimated); Status verified 2012-02

CONDITIONS: Children; Malnutrition
Keywords: SAM; RUTF; BIA; D2O; Children with severe malnutrition
MeSH Terms: conditions — Malnutrition | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): Parent/care givers of children with severe malnutrition in enrolled in this group will be given nutrition education using the principles of infant and young child feeding (IYCF) and dietary diversification
  Interventions: Behavioral: Nutrition education
- Group 2 (Active Comparator): Ready to use therapeutic food (RUTF / PlumpyNut)will be provided to parent/care givers of children with severe malnutrition in enrolled in this group
  Interventions: Dietary Supplement: RUTF

INTERVENTIONS:
Behavioral: Nutrition education — Parent/care givers of children with severe malnutrition in enrolled in this group will be given nutrition education using the principles of infant and young child feeding (IYCF) and dietary diversification
  Arms: Group 1
Dietary Supplement: RUTF — Ready to use therapeutic food (RUTF / PlumpyNut) will be provided to the parent/care givers of children with severe malnutrition in enrolled in this group
  Arms: Group 2

SUMMARY:
This project is being conducted with an aim to find out energy expenditure, body composition and recovery rates in children with severe acute malnutrition (SAM) receiving community-based nutritional rehabilitation therapy

DETAILED DESCRIPTION:
Objectives

1. To assess energy expenditure and body composition by stable isotope techniques in children with Severe Acute Malnutrition
2. To evaluate the potential usefulness of body composition assessment as a predictor of outcome in children with SAM, based on stable isotope technique and multi-frequency bioelectrical impedance analysis (BIA)

Inclusion criteria

* Parents of children of age 6 months to 3 years
* Resident of study area

Exclusion criteria

* Children with congenital malformations
* Chronic debilitating illnesses
* Refusal by parents to enroll in study

ELIGIBILITY:
Inclusion Criteria:

* Parents of children of age 6 months to 3 years
* Resident of study area

Exclusion Criteria:

* Children with congenital malformations
* Chronic debilitating illnesses
* Refusal by parents to enroll in study

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2010-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Body composition | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zulfiqar A Bhutta, MBBS,FCPS,FRCP,PhD, Principal Investigator — Aga Khan University
Locations (2):
- Pakistan (2):
  - Aga Khan Univeristy, Karachi, Sindh
  - Aga Khan University, Karachi, Sindh